CLINICAL TRIAL: NCT02017652
Title: Validation of FORE-SIGHT Cerebral & Tissue Oximeter to Measure Cerebral & Somatic Tissue Oxygen Saturation Measurements at Different Body Locations on Neonates ≤ 5 kg
Brief Title: Validation of Fore-Sight Cerebral & Tissue Oximeter Saturation Measurements on Neonates ≤ 5 kg
Acronym: FORE-SIGHT
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Other Study IDs: FORE-SIGHT
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Bowel Motility
Keywords: bowel motility; cerebral perfusion; intestinal perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm Infants: Preterm infants 32 to 36 weeks will be eligible for this study

SUMMARY:
CASMED, INC. wishes to validate the next generation FORE-SIGHT-II (FS-II) NIRS tissue oximeter monitor for neonatal brain and somatic tissue oxygen saturation (StO2) measurements. This monitor was recently FDA cleared for use on adult subjects.

DETAILED DESCRIPTION:
1. Validate FS-II abdominal StO2 measurements from the intestines, liver, and flank to umbilical venous and arterial blood oxygen saturation.
2. Validate FS-II cerebral StO2 measurements against the predicate FDA cleared FORE-SIGHT-I (FS-I) monitor.
3. Collect data from FS-II sensors on the forehead and abdomen (intestine) for 24 hours to compare dynamic changes vs the pulse oximeter. For larger neonates, add a predicate FS-I sensor to the opposite side forehead for dynamic comparison to FS-II measurements.
4. Obtain abdominal Near Infrared Spectroscopy (NIRS) data simultaneous with accepted measures of bowel motility (a. frequency and composition of stools, and b. Ultrasound assessment for the frequency and magnitude of bowel peristalsis, if available).

ELIGIBILITY:
Inclusion Criteria:

Neonatal subjects (32 to 36 and 6/7 weeks), with umbilical venous catheterization will be enrolled from the Neonatal Intensive Care Unit.

Exclusion Criteria:

Enrollment in other studies during study period. Inability to tolerate ultrasounds or NIRS sensors

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal subjects (32 to 36 and 6/7 weeks), with umbilical venous catheterization will be enrolled from the NICU. Demographic information of the subject will be recorded, including race, gender, weight, gestational age (GA), study age, and diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
StO2 measurement from intestines, liver and flank at time of venous and arterial blood oxygen saturation. | 1 hour
  At or immediately following an umbilical venous blood draw for CO-oximetry, the FS-II NIRS Small sensor will be briefly placed on the abdominal wall for spot check measurements over the 1) left & 2) right flank, 3) liver and on three intestine locations: just inferior and lateral to the umbilicus in the 4) Right Lower Quadrant (RLQ) and 5) Left Lower Quadrant (LLQ) positions, as well as 6) Mid Lower Quadrant (MLQ). Then a reference FS-I measurement of the 7) flank for 2 minutes will be done.
Cerebral StO2 measurements from Fore-Sight FS-II monitor and Fore-Sight-I (FS-I) monitor. | 1 hour
  Following abdominal measurements, the FS-II Small sensor will be placed on the head with the following positions in the following sequence 1) forehead, over the frontal cortex for two minutes; 2) the FS-II sensor is lifted off the head and placed back in the same forehead position to make a repeat measurement for two minutes; and 3) on the side of the head above the ear (frontal and parietal cortex) for two minutes. For reference cerebral measurements, a FDA cleared FS-I Small sensor will be placed on the 4) forehead for two minutes; 5) the FS-I sensor will be removed and replaced on the same forehead position to make a repeat measurement for two minutes. The sensors will take a measurement of 2 minutes in each position and 10 minutes total.
Pulse and Tissue oxygen saturation and infant activity | 24 hours
  Then two FS-II Small sensors will be attached longer term, one sensor on the forehead and one sensor on the abdomen (RLQ), with neonatal adhesives to allow monitoring for up to 24 hours. Dynamic changes of StO2 at these locations will be observed, along with pulse oximetry SpO2 to capture any acute events such as apnea and bradycardia, which will help in modeling and verifying dynamic StO2 change behavior within the FS-II algorithm. FS-II, and pulse oximetry data will be collected simultaneously on a laptop computer.
Stool Interference Index over 24 hrs. | 24 hours
  To calculate abdominal StO2 over the intestine regions, FORE-SIGHT also measures a stool interference index, which is used to compensate the algorithm to calculate StO2 correctly. This stool interference index is hypothesized to be also useful as a bowel motility index based on its variability over time. To test this hypothesis, the following two references for bowel motility will be tested: a) the study site will minimally record the number of stools for a period up to 24 hours. The event field in the laptop computer will be used to note each observation. b) if the study site has the capacity, abdominal ultrasound will be used to observe for the frequency and magnitude of bowel peristalsis. These impressions will be added to an event field in the laptop computer.

CONTACTS AND LOCATIONS:
Overall Officials: Anuup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States